CLINICAL TRIAL: NCT04424940
Title: TOMEKA® Project Was Sponsored by the University of Kinshasa: it's an Observational Study by Its Reviewed Documentation
Brief Title: COVID-19 Lessons Learned: the Outcome of TOMEKA® Project is to Teach
Acronym: MD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Kinshasa (Other)
Collaborators: University Ghent (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Guyguy K Tshima, MD, Principal Investigator, University of Kinshasa
Other Study IDs: UKinshasa; Tshima Guyguy Kabundi (Other: University of Kinshasa)
Record Dates: First submitted 2020-05-20; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: TOMEKA®; Treatment; COVID-19; Education
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Living in Canada and being health-worker in the first line face to COVID-19, investigator outcome is to teach an experience or explain the disease using a review and get people prepared to COVID-19 treatment focused on adherence to the HIV approved 2006-2007 protocol at Ghent University but the review shows an older different study approved at the University of Kinshasa and its ethics approval that again is an old document. So no ethics document supporting the study exists as it is now and no registration. It is an observational study and therefore would not usually require registration in order for the results to be published. It is not a type of secondary literature. The formula TOMEKA® (Mix porridge of maize, sorghum, and soya) follows FOOD + HEALTH CLAIM. It is scientifically justified, relevantly used, and correctly communicated. Methodology: sufficient data? scientific consensus? correct methodology? correct population? context: significant results? context of use, realistic ingestion? correct target group? communication: consumer perception? exaggerated/insinuative, clear, precise, complete, correct information? not misleading? correctly presented? The product TOMEKA® tried to fulfill to above questions in a fitting way with COVID-19 which is an emerging, rapidly evolving situation without a vaccine.

DETAILED DESCRIPTION:
On 12/06/2020 worldwide, COVID-19 affected 7 273 958 confirmed cases with 413 372 deaths, 97 894 confirmed in Canada with 8 048 deaths, 53 666 confirmed cases in Quebec with 5 148 deaths, 4 637 confirmed cases with 101 deaths in the Democratic Republic of the Congo where the situation is disastrous: an immense country and the ways of communication are difficult and damaged. It becomes gymnastics to get a drug package.

The principal investigator provide the details of this study to be available to the public in getting knowledge of Covid-19 and micronutrients using the product TOMEKA®.

The individual contribution of ingredients in the nutritional composition of TOMEKA® (mixed flour). Composition of TOMEKA® (Clinical Research Protocol): 100 g of TOMEKA contain 20.1 g of protein; 57.8 g of carbohydrates, 10.1 g of lipids; 8.5 mg iron; 117.6 mg Calcium; 16.6 mg Sodium; 55 μg of Selenium and 378.6 kcal of energy.TOMEKA will be made with soy, maize, sorghum. The above calculations were made with the food composition table (no laboratory analyzes).

Quantity to be served per meal (in g): 30 g for 6-8 months (113,4 Kcal of Energy per served meal). 40 g for 9-11 months (151 Kcal): 50 g for 12-23 months and more expecting to provide 189 Kcal of energy per served per meal. Each group needs 4-5 meals a day to get the equivalent of their daily nutritional needs.

The study will focus on Selenium, a powerful non-enzymatic antioxidant, more powerful than Vit C and Vit E combined. The formula TOMEKA® follows FOOD + HEALTH CLAIM.

A clear device to follow micronutrients and Covid-19 symptoms:

Example 1: Vitamin D and Covid-19 (Press release from the National Academy of Medicine in France May 22, 2020) Vitamin D is a prohormone synthesized in the dermis under the effect of ultraviolet rays, that is to say of the rays of the sun, then transported in the liver and the kidney where it is transformed into an active hormone. It is responsible for the intestinal absorption of calcium and bone health, but vitamin D also has unconventional effects. In particular, it modulates the functioning of the immune system by stimulating macrophages and dendritic cells [1,2,3]. It plays a role in regulating and suppressing the cytokine inflammatory response which causes acute respiratory distress syndrome which characterizes the severe and often lethal forms of Covid-19. A significant correlation between low serum vitamin D levels and mortality by Covid-19 has been shown [4]. This phenomenon generally follows a North-South gradient, although there are exceptions such as the Nordic countries where the supplementation of the nutrients in vitamin D, in particular milk products, is systematic. On the other hand, the countries of southern Europe surprisingly display a high prevalence of vitamin D deficiency despite higher sunshine [5]. This would explain why children who receive vitamin D regularly have asymptomatic forms of Covid-19 and fewer complications. Vitamin D cannot be considered as a preventive or curative treatment for SARS-CoV-2 infection; but by mitigating the inflammatory storm and its consequences, it could be considered as an adjunct to any form of therapy.

The National Academy of Medicine in France recalls that the administration of vitamin D orally is a simple, inexpensive measure and reimbursed by Health Insurance; - confirms its recommendation to ensure vitamin D supplementation in the French population in a report in 2012 [2]; - recommend that the serum vitamin D level (i.e. 25OHD) be measured quickly in people over 60 years of age with Covid-19 and that it be administered in the event of a deficiency, a loading dose of 50,000 to 100,000 IU which could help limit respiratory complications; - recommends providing vitamin D supplementation of 800 to 1,000 IU / day in people under the age of 60 as soon as the diagnosis of Covid-19 is confirmed.

Example 2: Selenium and Covid-19

Now is the time to give extra attention to a balanced diet and assure an optimum dietary micronutrient and vitamin intake! Particularly the micronutrient selenium plays an essential role in antioxidant functioning and helps to alleviate the negative health impacts of viral infections, including inflammation of the lungs (see e.g. https://lnkd.in/eqAGhDH).

Particularly elderly people are often selenium-deficient, which was proven to be the case in e.g. Italy (see https://lnkd.in/epFKVEY). However, when taking micronutrient and vitamin supplements, also follow the instructions to avoid over-supplementation! A healthy and balanced diet is the safest way towards an appropriate dietary micronutrient and vitamin intake.

Description of what investigators will measure:

1. The Production of Medical Knowledge:
2. Learning medicine:

How it will be measured:

1. The Production of Medical Knowledge: Anthropology/Medicine. It is substantial and it showed by the title.
2. Learning medicine: The clinical trial shows that medical anthropology connects anthropology and social theory generally with some of the more significant questions of our epoch with the COVID-19 pandemic.

And at what time points it will be measured:

1. The Production of Medical Knowledge: the principal investigator has received notifications from Researchgate about 700 researchers who read his research theme, so it deserves to be widely read and taught.
2. Learning medicine: This is an original trial, which combines theoretical argument with empirical observation

Objectives:

1. Investigators would like the participant to accept the notion that all knowledge is socially and culturally constructed.
2. Investigators would examine the contexts in which that knowledge is produced talking on the theme of nutrition in research and aiming to act in medicine, psychiatry, epidemiology, and anthropology.
3. Investigators would like the participant acts in behavioral medicine, public health, epidemiology, anthropology as well as .nutrition.

The hypothesis of investigators work:

1. Patients with COVID-19 have an increased demand for Selenium
2. Selenium supplementation reduces the viral rate
3. Selenium supplementation improves the BMI of COVID-19 patients
4. Selenium supplementation reduces COVID-19 related morbidity
5. Selenium supplementation postponed COVID-19 related mortality
6. Selenium supplementation is adjuncted to any form of COVID-19 therapy with nutrition education
7. Nutrition education improves health status
8. Selenium supplementation and nutrition education should be incorporated into the global Nutritional care and support of COVID-19 patients

   Methodology: observational study using a questionnaire.

   Study Population:

   Age: 15-75

   Sex: M, F

   Inclusion Criteria:

   Fulfill Inclusion criteria and accept:

   The participant is asked on the symptoms of the COVID-19 with a questionnaire. If he/she can write yes to any of these questions in order to be tested:

   In the past 4 hours, have you taken any medicines for fever or headaches, such as acetaminophen (Paracetamol, Tylenol, Tempra), ibuprofen (Advil, Motrin) or Aspirin?

   Yes

   No

   Do you have a thermometer to take your body temperature?

   Yes

   No

   If you don't have a thermometer, do you have any of the following symptoms: warm forehead, muscle or joint pain, chills, general weakness?

   Yes

   No

   In the past 24 hours, have you had trouble breathing or been short of breath?

   Yes

   No

   In the past 24 hours, have you had chest pain?

   Yes

   No

   Do you have a cough? Or if you have a health condition that is causing you to cough, is your cough worse than usual?

   Yes

   No

   In the past 24 hours, have you had a sore throat?

   Yes

   No

   In the past 24 hours, have you had a runny nose?

   Yes

   No

   In the past 24 hours, have you felt a loss of smell (in the absence of nasal congestion)?

   Yes

   No

   In the past 24 hours, have you had diarrhea (three or more bowel movements)?

   Yes

   No

   In the past 24 hours, have you had a headache?

   Yes

   No

   In the past 24 hours, have you felt more tired than usual and unable to carry out your daily activities?

   Yes

   No

   COVID-19 patients confirmed

   be regular on appointments

   Exclusion Criteria:

   COVID-19 suspected clinically

   Children

   refuse to participate

   Initial assessment for the exclusion of suspected Covid-19 cases:

   - New or exacerbated cough: Yes/No

   - Sore throat: Yes/No

   - Fever: Yes/No

   - Intestinal gastritis symptoms (Diarrhea, nausea or vomiting): Yes/No

   - Anosmia (loss of smell) / Ageusia (loss of taste): Yes/No
   * Shortness of breath: Yes/No
   * Sputum production: Yes/No
   * Weakness: Yes/No
   * Headache: Yes/No
   * Myalgia / athralgia: Yes/No
   * Nasal congestion: Yes/No
   * Hemoptysis: Yes/No
   * Conjunctivitis: Yes/No

   Comments:

   If yes to any of these questions: rule out an acute health condition. If no acute cause identified, consider the person as a probable case and transfer to the warm unit.

2. Atypical geriatric signs

* Sudden loss of autonomy (less than 1 week)
* Sudden change in mental state (over 1 week)
* Sudden change in behavior (new behavior or cessation of behavior (less than 1 week)
* Geriatric fever (Oral or rectal temperature greater than or equal to 37.8 C or if increase of 1.1 C compared to the usual normal T)

Other comments:

………………………………………………………………………………………………………….. ........................................................................................................................................................................................................................................................................................................................................................................................................................................................

3. Physical examination inspection:

* Assessment of mental state
* Attention span: attentive, not attentive
* State of consciousness: hyper-alert (or agitation), Lethargic (verbal), alert stupor (physical, comatose

  4. Basic settings:

Vital signs:

Pulse: ……… / min TA: .......... / ……………. T: ................ C (fever if bu oral or rectal sup or equal 37.8 C or if 1.1 C increase compared to the usual normal T)

Breathing:

Frequency: ......... / min

Type: Abdominal chest

Amplitude: normal deep surface

Rhythm: regular irregular

Draw: yes no

Saturation (normal to 94% and +, unless otherwise indicated):

Saturation: ............% ambient AIr With O2 …… ..L / min

5. Auscultation:

Anterior side

Abnormal noise: Yes No

Name if possible:

Sibilant

Ronchis

Right bronchus (A)

Left bronchus (B)

Posterior side

Presence of abnormal noise:

Yes

No

Name if possible:

Sibilant

Crackling

Lower right row

Left lower lobe

6. Medical decision making

Prescribed screening test (oro-nasopharyngeal sample): yes no

If the sample confirms the presence of COVID-19, isolate the patient in the warm unit.

7. Clinical monitoring of COVID-19 confirmed or suspected

Stable patient

Respiratory rate : q 2h and as needed

SpO2 and Temperature: per day and as needed

Blood pressure and Cardiac frequency: per day

Unstable patient (having had an episode of respiratory distress)

Respiratory rate: every hour and as needed

SpO2 and Temperature: per day and as needed

Surname and first name of doctor

Permits

Signature

DD / MM / YYYY

HH: MM

References:

1. - Liu PT, Stenger S, et al. Toll like receptor triggering of a vitamin D mediated humanantimicrobial response. Science, 2006, 311 : 1770.
2. - Rapport de l'Académie nationale de médecine. Statut vitaminique, rôle extra osseux etbesoins quotidiens en vitamine D. Bull Acad Natle Med. 2012, 196, 1011.
3. - Laird E, Rhodes JM and Kenny RA. Vitamin D and inflammation : potential implications for severity of Covid-19. Irish med J, 2020, 113 : 81.
4. - McCartney DM, Byrne DG. Optimisation of vitamin D status impact mortality fromSARS -CoV-2 infection Irish Med J .2020 113 : 58.5- Lips P, Cashman KD, et al. Current vitamin D status in European and Middle East countries and strategies to prevent vitamin D deficiency : a position statement of the European Calcified Tissue Society. Eur J Endocrinol, 2019, 180 : P23-P54.

Links:

https://lnkd.in/eqAGhDH https://lnkd.in/epFKVEY

ELIGIBILITY:
Inclusion Criteria:

* Fulfill Inclusion criteria and accept
* COVID-19 patients confirmed
* be regular on appointments

Exclusion Criteria:

* COVID-19 suspected clinically
* Children
* refuse to participate

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Age: 15-75
  * Sex: M, F
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-TOMEKA® usage as assessed by Education | 9 months
  Change people's behaviour

SECONDARY OUTCOMES:
Change From Baseline in nutraceuticals usage on the care of the Covid-19 at 9 months | 9 months
  Change people's behaviour

CONTACTS AND LOCATIONS:
Overall Officials: GUYGUY KABUNDI TSHIMA, MD, Principal Investigator — University of Kinshasa
Locations (1):
- Cliniques Universitaires de Kinshasa, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Through researchgate website
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the beginning of the study and follow-up
Access Criteria: for free
URL: https://www.researchgate.net/publication/319997498_A_prospective_study_on_weight_evolution_of_people_living_with_HIV-AIDS_under_antiretroviral_drugs_in_malaria_endemic_areas

REFERENCES:
- [Background] This phenomenon generally follows a North-South gradient, although there are exceptions such as the Nordic countries where the supplementation of the nutrients in vitamin D, in particular milk products, is systematic. On the other hand, the countries of southern Europe surprisingly display a high prevalence of vitamin D deficiency despite higher sunshine
- [Background] This would explain why children who receive vitamin D regularly have asymptomatic forms of Covid-19 and fewer complications. Vitamin D cannot be considered as a preventive or curative treatment for SARS-CoV-2 infection; but by mitigating the inflammatory storm and its consequences, it could be considered as an adjunct to any form of therapy.
- [Background] The National Academy of Medicine in France recalls that the administration of vitamin D orally is a simple, inexpensive measure and reimbursed by Health Insurance; - confirms its recommendation to ensure vitamin D supplementation in the French population in a report in 2012 [2]; - recommend that the serum vitamin D level (i.e. 25OHD) be measured quickly in people over 60 years of age with Covid-19, and that it be administered in the event of a deficiency , a loading dose of 50,000 to 100,000 IU which could help limit respiratory complications; - recommends providing vitamin D supplementation of 800 to 1,000 IU / day in people under the age of 60 as soon as the diagnosis of Covid-19 is confirmed.
- [Result] Now is the time to give extra attention to a balanced diet and assure an optimum dietary micronutrient and vitamin intake! Particularly the micronutrient selenium plays an essential role in antioxidant functioning and helps to alleviate negative health impacts of viral infections, including inflammation of the lungs
- [Result] Particularly elderly people are often selenium-deficient, which was proven to be the case in e.g. Italy
- [Result] However, when taking micronutrient and vitamin supplements, also follow the instructions to avoid over-supplementation! A healthy and balanced diet is the safest way towards an appropriate dietary micronutrient and vitamin intake.
- [Result] Vitamin D is a prohormone synthesized in the dermis under the effect of ultraviolet rays, that is to say of the rays of the sun, then transported in the liver and the kidney where it is transformed into an active hormone. It is responsible for the intestinal absorption of calcium and bone health, but vitamin D also has unconventional effects. In particular, it modulates the functioning of the immune system by stimulating macrophages and dendritic cells.
- [Result] It plays a role in regulating and suppressing the cytokine inflammatory response which causes acute respiratory distress syndrome which characterizes the severe and often lethal forms of Covid-19. A significant correlation between low serum vitamin D levels and mortality by Covid-19 has been shown.
- See also: Guillin OM, Vindry C, Ohlmann T, Chavatte L. Selenium, Selenoproteins and Viral Infection. Nutrients. 2019;11(9):2101. Published 2019 Sep 4. doi:10.3390/nu11092101 — https://lnkd.in/eqAGhDH
- See also: Lauretani F, Semba RD, Bandinelli S, et al. Low plasma selenium concentrations and mortality among older community-dwelling adults: the InCHIANTI Study. Aging Clin Exp Res. 2008;20(2):153-158. doi:10.1007/BF03324762 — https://lnkd.in/epFKVEY